CLINICAL TRIAL: NCT00648973
Title: Evaluation of Nasal Congestion Clinical Efficacy for Diphenhydramine 25 mg and Diphenhydramine 50 mg in Seasonal Allergic Rhinitis: a Randomized, Double-blind, Placebo and Pseudoephedrine Controlled Study
Brief Title: To Determine if Diphenhydramine Works for Nasal Congestion at Two Different Doses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2341002
Record Dates: First submitted 2008-03-20; First posted 2008-04-01 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Nasal Congestion
Keywords: Seasonal Allergic Rhinitis, nasal congestion
MeSH Terms: conditions — Nasal Obstruction; Rhinitis, Allergic, Seasonal | interventions — Diphenhydramine; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Diphenhydramine 50 mg
  Interventions: Drug: Diphenhydramine 50 mg
- 2 (Experimental): Diphenhydramine 25 mg
  Interventions: Drug: Diphenhydramine 25 mg
- 3 (Active Comparator): Pseudoephedrine 120 mg
  Interventions: Drug: Pseudoephedrine 120 mg

INTERVENTIONS:
Drug: Diphenhydramine 50 mg — Three times daily: two diphenhydramine 25 mg capsules
  Twice daily: one pseudoephedrine-matching placebo tablet
  Other Names: Active: Lot # 070PB6 Formula # W015990-0002
  Arms: 1
Drug: Diphenhydramine 25 mg — Three times daily: one diphenhydramine 25 mg capsule and one diphenhydramine-matching placebo capsule
  Twice daily: one pseudoephedrine-matching placebo tablet
  Other Names: Active: Lot # 070PB6 Formula # W015990-0002
  Arms: 2
Drug: Pseudoephedrine 120 mg — Three times daily: two diphenhydramine-matching placebo capsules
  Twice daily: one pseudoephedrine 120 mg tablet
  Other Names: Active: Lot # INT-06-115 Formula # W015721-0004
  Arms: 3

SUMMARY:
The study was to determine if the drug worked to relieve nasal congestion experienced by people with seasonal allergies.

DETAILED DESCRIPTION:
Subjects who met the inclusion/exclusion criteria were enrolled into the placebo run-in phase of the study on Day -7 (prerandomization, Visit 1). Baseline symptom scores were established during this run-in phase.

Subjects with moderate nasal congestion who took at least 80% of their study medication during the run-in phase were eligible for enrollment in the two-week double-blind phase of the study and were randomized on Day 1 (randomization, Visit 2). They were treated for two weeks with their assigned medication. The severity of signs/symptoms were evaluated by the subjects every morning and night and by the investigator at each visit on Day 7 and Day 14.

In addition, the subject and investigator provided a global evaluation of response to treatment on Day 7 and Day 14. Safety was evaluated by adverse events reported during the study, vital signs, and the incidence of somnolence.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy males and females
* 12 to 65 years of age
* hypersensitivity to specific pollens for a minimum of 2 years prior to study start
* appropriate SAR sign/symptoms scores

Exclusion Criteria:

* pregnancy, lactation and contraception issues
* contraindicated medications or therapies
* evidence of clinical, dietary, lifestyle or psychiatric issues, which in the opinion of the investigator, could increase the risk to the subject or research staff, or interfere with the interpretation of study results

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the subject's mean reflective nasal congestion/stuffiness symptom score | every 12-hours over the 14-day treatment period

SECONDARY OUTCOMES:
Change from baseline in the subject's mean reflective Total Nasal Symptom (TNS) Score | 14 Days
Change from baseline in the subject's mean instantaneous TNS Score | 14 Days
Change from baseline in the subject's mean reflective Total SAR Symptom (TSS) Score | 14 Days
Change from baseline in the subject's mean instantaneous TSS Score | 14 Days
Change from baseline in the subject's mean reflective score for each of the seven remaining individual SAR symptoms, excluding nasal congestion/stuffiness | 14 Days
Change from baseline in the subject's mean instantaneous score for each of the eight individual SAR symptoms | 14 Days
Onset of action for diphenhydramine treatment for nasal congestion/stuffiness was determined by comparing the change from baseline in the subject's instantaneous nasal congestion/stuffiness scores for diphenhydramine versus placebo | taken at 15, 30, 60 and 90 minutes after the initial dose. Baseline was the score taken just prior to the initial dose.
Onset of action for diphenhydramine treatment for allergic rhinitis symptoms was determined by comparing the change from baseline in the subject's instantaneous TNS scores for diphenhydramine versus placebo | taken at 15, 30, 60 and 90 minutes after the initial dose. Baseline was the score taken just prior to the initial dose
Duration of action for diphenhydramine for treatment of nasal congestion/stuffiness was evaluated by comparing the change from baseline in the subject's mean instantaneous nasal congestion/stuffiness scores for diphenhydramine versus placebo | taken at the six-hour trough (just prior to the 8:00 pm dose) and the 12-hour trough (just prior to the 8:00 am dose)
Duration of action for diphenhydramine for treatment of allergic rhinitis symptoms was evaluated by comparing the change from baseline in the subject's mean instantaneous TNS scores for diphenhydramine versus placebo | taken at the six-hour trough (just prior to the 8:00 pm dose) and the 12-hour trough (just prior to the 8:00 am dose)
Time to maximal effect was assessed by a by-day analysis of the primary efficacy endpoint and select secondary endpoints | 14 Days
Subject's global evaluation of response to treatment | at Visits 3 and 4, analyzed separately at each visit
Change from baseline in the Investigator's TNS score | at Visits 3 and 4, analyzed separately for each visit. Baseline was the score at Visit 1
Change from baseline in the Investigator's TSS score | at Visits 3 and 4, analyzed separately for each visit. Baseline was the score at Visit 1
Change from baseline for each of the eight individual Investigator's SAR symptoms | at Visits 3 and 4, analyzed separately for each visit. Baseline was the score at Visit 1
Investigator's global evaluation of the subject's response to treatment | at Visits 3 and 4, analyzed separately for each visit
Number and percentage of subjects experiencing adverse events | Duration of study
Change from baseline and potentially clinically important vital signs (systolic and diastolic blood pressure, pulse, and respiratory rate) | Duration of study
Occurrence of somnolence | Overall and weekly

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Israel, BS, Study Director — McNeil Consumer Healthcare Division of Mc-Neil-PPC, Inc.
Locations (12):
- United States (12):
  - Benchmark Research - Austin, Austin, Texas
  - Allergy and Asthma Associates, Austin, Texas
  - Lovelace Scientific Resources, Austin, Texas
  - Allergy/Immunology Research Center of North Texas, Dallas, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Benchmark Research - San Angelo, San Angelo, Texas
  - Sun Research Institute, San Antonio, Texas
  - Biogenics Research Institute, San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas